CLINICAL TRIAL: NCT02776163
Title: Postoperative Concurrent Chemoradiotherapy in Treating Patients With High-Risk Salivary Gland Carcinomas of Head and Neck, A Non-Randomized, Phase II Trial
Brief Title: Postoperative Concurrent Chemoradiotherapy in Treating Patients With High-Risk Salivary Gland Carcinomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Guopei Zhu, M.D., Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016HNRT002
Record Dates: First submitted 2016-05-12; First posted 2016-05-18 (Estimated); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Salivary Gland Tumors; Head and Neck Cancer
Keywords: Salivary Gland Tumors; Head-an-Neck cancer; Concurrent Chemoradiotherapy; High-Risk; Cisplatin; Docetaxel
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — nedaplatin; Docetaxel; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACC (Experimental): Intensity-modulated radiotherapy+concurrent chemotherapy with docetaxel and Nedaplatin
  Interventions: Drug: Nedaplatin; Drug: Docetaxel; Radiation: Intensity-modulated radiotherapy
- Non-ACC (Experimental): Intensity-modulated radiotherapy+concurrent chemotherapy with docetaxel and Nedaplatin
  Interventions: Drug: Nedaplatin; Drug: Docetaxel; Radiation: Intensity-modulated radiotherapy

INTERVENTIONS:
Drug: Nedaplatin — nedaplatin 35mg/m^2，D1-2，2 cycles
Drug: Docetaxel — Docetaxel 70mg/m^2，D1，2 cycles
Radiation: Intensity-modulated radiotherapy — a total dose of 60-66Gy in 30-33 fractions over 6-7 weeks

SUMMARY:
This is a non-randomized, phase II, open label study of postoperative current chemoradiotherapy for high-risk malignant salivary gland tumors of head and neck.The primary purpose of this study is to evaluate the efficacy and safety of concurrent chemoradiotherapy in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven diagnosis of a malignant salivary gland tumor of intermediate or high-grade
2. Pathologic stage T3-4 or N1-3 or T1-2, N0 with a close (≤ 5mm) or microscopically positive surgical margin
3. Surgical resection with curative intent within 8 weeks prior to registration, with no evidence of gross tumor residual
4. No evidence of distant metastases
5. No synchronous or concurrent head and neck primary tumors
6. Karnofsky score over 60
7. Adequate organ function including the following:

   1. Absolute neutrophil count (ANC) >= 1.5 * 10^9/l
   2. Platelets count >= 100 * 10^9/l
   3. Hemoglobin >= 10 g/dl
   4. AST and ALT <= 2.5 times institutional upper limit of normal (ULN)
   5. Total bilirubin <= 1.5 times institutional ULN
   6. Creatinine clearance >= 50 ml/min
   7. Serum creatine <= 1 times ULN
8. Signed written informed consent

Exclusion Criteria:

1. Evidence of distant metastasis
2. Prior chemotherapy or anti-cancer biologic therapy for any type of cancer, or prior radiotherapy to the head and neck region
3. Other previous cancer, except for in situ cervical cancer and cutaneous basal cell carcinoma
4. Pregnant or breast-feeding females, or females and males of childbearing potential not taking adequate contraceptive measures
5. Presence of an uncontrolled concomitant illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 2 years
  from date of enrollment until date of first documented disease progression or death from any cause, assessed up to 2 years

SECONDARY OUTCOMES:
Overall survival rate | 2 years
  from date of enrollment until date of first death from any cause, assessed up to 2 years
Acute toxicity profiles, graded according to the NCI CTCAE version 3.0 | up to 6 weeks
  Number of participants with treatment-related acute toxicity as assessed weekly by CTCAE v3.0 during the course of treatment
Late toxicity profiles, graded according to the NCI CTCAE version 3.0 | up to 2 years
  Number of participants with treatment-related late toxicity as assessed every 3 months by CTCAE v3.0 up to 2 years
Score of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck Core 35 (EORTC QLQ-HN35) during the concurrent treatment | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
  QoL score will be documented on each weekend during the course of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Guopei Zhu, M.D., Principal Investigator — Shanghai Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai ninth people's hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No